CLINICAL TRIAL: NCT03444090
Title: Impacts of Inspection During Instrument Insertion on Colonoscopy Quality: a Prospective Randomized Controlled Trial
Brief Title: Impacts of Inspection During Instrument Insertion on Colonoscopy Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evergreen General Hospital, Taiwan (Other)
Responsible Party: Principal Investigator, Chi-Liang Cheng, Director of Gastroenterology, Evergreen General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EGH-2017-1
Record Dates: First submitted 2018-02-10; First posted 2018-02-23 (Actual); Results first posted 2019-05-09 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-02

CONDITIONS: Colon Polyp; Colon Adenoma
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insertion/withdrawal colon polypectomy (Experimental): For participants assigned in the experimental group, the colon is washed and the debris is suctioned as the colonoscopy is slowly inserted from rectum to cecum. Deliberate and systematic inspection of the mucosa is performed with adequate insufflation during both insertion and withdrawal phases.Colon polypectomy for polyp size <10 mm will be performed when they are identified during insertion and withdrawal of the colonoscope. Colon polypectomy for polyp size >10 mm will be performed only during withdrawal of the scope.
  Interventions: Procedure: Colon polypectomy
- Withdrawal colon polypectomy (Active Comparator): For participants assigned in the control group, deliberate mucosa inspection and colon polypectomy will be performed exclusively on colonoscopy withdrawal.During insertion, minimal mucosal inspection and insufflation are applied to efficiently advance the instrument into cecum.
  Interventions: Procedure: Colon polypectomy

INTERVENTIONS:
Procedure: Colon polypectomy — For participants assigned into the experimental group, colon lumen is washed and the debris is suctioned as the colonoscopy is slowly inserted from rectum to cecum. Deliberate and systematic inspection of the mucosa is performed with adequate insufflation during both the insertion and withdrawal phases. Colon polyps with size <10 mm are removed as they are identified on insertion and withdrawal. Polyps with size >10 mm are removed only during withdrawal.
  For participants assigned into the control group, deliberate inspection and polyp removal are performed exclusively on colonoscopy withdrawal.During insertion, minimal mucosal inspection and insufflation are applied to efficiently advance the instrument into cecum.

SUMMARY:
Small colon polyps which are found during colonoscopy insertion are sometimes difficult to find during withdrawal and thus missed. The investigators aim to evaluate the differences of colon polyp/adenoma detection rates of patients undergoing additional inspection and polypectomy during insertion as compared to the patients undergoing traditional practice of careful inspection and polypectomy performed entirely during withdrawal of colonoscopy.

DETAILED DESCRIPTION:
Participants will be randomly assigned by a research assistant, by using a computer-generated randomization sequence to undergo colonoscopy with either inspection and polypectomy during both insertion and withdrawal of colonoscope (study group) or inspection and polypecotmy entirely during withdrawal of colonoscope (control group). Randomization will be done via concealed allocation with a sealed envelope that designate study group or control group.

Colonoscopies will be performed by two experienced investigators by using a standard colonoscopy (CF-Q260AI or CF-Q260AL; Olympus Medical Systems Corp., Tokyo, Japan). All procedures are performed under moderate conscious sedation with fentanyl (United Biomedical, Taipei, Taiwan) and midazolam (Dormicum; Roche Pharmaceuticals, Basel, Switzerland) according to the current guidelines. Carbon dioxide insufflation is used for all endoscopic procedures. All participants receive 3-L polyethylene glycol (PEG; Klean-Prep, Helsinn Birex Pharmaceuticals Ltd., Dublin, Ireland) for bowel preparation. A split-dose of the PEG preparation is provided. The level of colon cleansing is prospectively evaluated with the Boston Bowel Preparation Scale score.

For participants assigned into the study group, the colonic lumen is washed with saline and the fluid and debris are suctioned as the instrument is slowly inserted from rectum to cecum. Deliberate and systematic inspection of the colonic mucosa is performed with adequate luminal insufflations during both the insertion and withdrawal phases. Polyp size is determined by comparison with open colonoscopic biopsy forceps pushed against the polyp or, in some cases of pedunculated polyp by direct measurement after retrieval. Polyps with size <10mm are removed as they are identified on insertion and withdrawal. Polyps with size ≥10mm are removed only during withdrawal.

For participants assigned into the control group, deliberate mucosal inspection and polyp removal are performed exclusively on instrument withdrawal. During insertion, minimal mucosal inspection and insufflation are applied to efficiently advance the instrument into cecum. If a polyp is found during insertion, investigators are instructed to make a mental note of it and find it during withdrawal for polypectomy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 45 years or older.
* Agree to participate the study and provide a written informed consent

Exclusion Criteria:

* Previous surgical resection of the colon or rectum
* Inflammatory bowel disease
* Polyposis syndrome
* Previously incomplete colonoscopy
* Obstructive lesions of colon
* Inadequate bowel preparation, defined as Boston Bowel Preparation Scale score of 0 or 1 in any colon segment
* Gastrointestinal bleeding
* Allergy to fentanyl or midazolam
* American Society of Anesthesiology classification of physical status 3 or higher
* Mental retardation
* Pregnancy
* Refusal to provide a written informed consent

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chiliang Cheng, Principal Investigator — Evergreen General Hospital
Locations (1):
- Evergreen General Hospital, Taoyuan District, Taiwan

REFERENCES:
- [Derived] Cheng CL, Kuo YL, Liu NJ, Tang JH, Fan JW, Lin CH, Tsui YN, Lee BP, Hung HL. Comparison of polyp detection during both insertion and withdrawal versus only withdrawal of colonoscopy: A prospective randomized trial. J Gastroenterol Hepatol. 2019 Aug;34(8):1377-1383. doi: 10.1111/jgh.14613. Epub 2019 Feb 27. PMID 30675926

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Insertion/Withdrawal Colon Polypectomy | Withdrawal Colon Polypectomy
Started | 214 | 214
Completed | 211 | 210
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insertion/Withdrawal Colon Polypectomy | Withdrawal Colon Polypectomy | Total
Number analyzed (Participants) | 211 | 210 | 421
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (8.5) | 58.2 (8.5) | 57.9 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 111 | 223
  Male | 99 | 99 | 198
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 211 | 210 | 421
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 211 | 210 | 421

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Detection of at Least One Adenoma Per Procedure
Description: Colon adenoma detection rate is defined as the proportion of colonoscopies where at least one adenoma is found.
Time Frame: During procedure, approximately one hour
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Insertion/Withdrawal Colon Polypectomy | Withdrawal Colon Polypectomy
Number analyzed (Participants) | 211 | 210
percentage of participants | 63.7 [56.6 to 70.0] | 68.1 [61.3 to 74.3]

2. Secondary Outcome: Mean Colon Adenoma Per Colonoscopy
Description: Mean colon adenoma per procedure is defined as the total number of adenomas detected divided by the number of colonoscopies.
Time Frame: During procedure, approximately one hour
Measure: Mean (Standard Deviation); unit: adenomas/colonoscopy
Arm/Group | Insertion/Withdrawal Colon Polypectomy | Withdrawal Colon Polypectomy
Number analyzed (Participants) | 211 | 210
adenomas/colonoscopy | 1.6 (2.0) | 1.9 (2.4)

ADVERSE EVENTS:
Time Frame: one month
Arm/Group | Insertion/Withdrawal Colon Polypectomy | Withdrawal Colon Polypectomy
All-Cause Mortality (participants affected / at risk) | 0/211 | 0/210
Serious Adverse Events (participants affected / at risk) | 0/211 | 0/210
Other Adverse Events (participants affected / at risk) | 0/211 | 0/210

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-07): https://cdn.clinicaltrials.gov/large-docs/90/NCT03444090/Prot_SAP_000.pdf